CLINICAL TRIAL: NCT00492349
Title: Varenicline Adjunctive Treatment in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, L. Elliot Hong, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00040322
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2017-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: Varenicline; Neurobiology; clinical trial; cognitive deficits; Schizophreniform Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Cognition Disorders | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Varenicline
  Interventions: Drug: Varenicline
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Varenicline 0.5mg po qd x 7 days then titrated to Varenicline 0.5mg po bid x 7 weeks
  Other Names: Chantix
  Arms: 1
Drug: Placebo — Placebo 0.5mg po qd x 7 days then titrated to Placebo 0.5mg po bid x 7 weeks
  Arms: 2

SUMMARY:
The principal aim of the project is to conduct an off-label adjunctive clinical trial evaluating varenicline as a treatment for core neurobiological and clinical deficits in schizophrenia, in addition to evaluating for smoking cessation in schizophrenia patients.

DETAILED DESCRIPTION:
This is a double-blind, placebo controlled clinical trial in schizophrenia patients. Outcome measures include biomarkers and clinical symptoms and functions, and smoking cessation. Neurobiological and cognitive markers will be measured for short term (2 weeks) and longer-term (8 weeks). Current schizophrenia treatments are mostly ineffective against primary negative symptoms and the cognitive and information processing deficits associated with the disorder. Previous research has identified several neurophysiological deficits in schizophrenia that are enduring, frequently occurring before psychosis, and mark the disease liability. These schizophrenia endophenotypes provide important targets for novel treatment development as they represent the core deficits of the disorder. We hypothesize that sustained nicotinic and dopaminergic modulation by varenicline may ameliorate the core neurobiological deficits seen in schizophrenia patients, which would lead to subsequent clinical improvement. Neurobiological and neurocognitive markers and clinical and functional measures will be obtained to determine 1) short-term effect of varenicline on biomarkers; and 2) longer-term improvement in clinical symptoms, smoking cessation, and functions; and how biomarker changes predict these improvements.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* DSM-IV Diagnosis of schizophrenia, schizoaffective disorder, or schizophreniform disorder
* Clinically stable with no change in antipsychotic medications and increase of daily dose for 4 weeks prior to enrollment
* Sufficient understanding of the study and risks (ESC score 10 or above)

Exclusion Criteria:

* Major medical illness history including, but not limited to, history of heart attack, stroke, TIA (transient ischemic attack)
* History of organic brain disorders that may affect neurophysiological measurements, including seizure disorder, brain tumor, head injury with evidence of significant cognitive deterioration
* DSM-IV diagnosis of substance dependence within 6 months except nicotine and marijuana
* On nicotine replacement therapy (nicotine patch, gum, or nasal spray)
* Uncontrolled blood pressure (persistent systolic above 155 or diastolic above 95)
* EKG of second or third degree atrioventricular (AV) block
* Renal insufficiency with estimated creatinine clearance <40 ml/min
* Women who have positive urine pregnancy tests
* Women who are pregnant, plan to become pregnant, or in breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2007-05; Primary Completion 2010-05 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L. Elliot Hong, M.D., Principal Investigator — Maryland Psychiatric Research Center, Department of Psychiatry, University of Maryland School of Medicine
Locations (3):
- United States (3):
  - UMB School of Medicine, Baltimore, Maryland
  - University of Maryland Medical System, Baltimore, Maryland
  - Maryland Psychiatric Research Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Hong LE, Thaker GK, McMahon RP, Summerfelt A, Rachbeisel J, Fuller RL, Wonodi I, Buchanan RW, Myers C, Heishman SJ, Yang J, Nye A. Effects of moderate-dose treatment with varenicline on neurobiological and cognitive biomarkers in smokers and nonsmokers with schizophrenia or schizoaffective disorder. Arch Gen Psychiatry. 2011 Dec;68(12):1195-206. doi: 10.1001/archgenpsychiatry.2011.83. Epub 2011 Aug 1. PMID 21810630
- See also: Click here for more information about the study: Varenicline Adjunctive Treatment in Schizophrenia — http://www.bioportfolio.com/resources/trial/98676/Varenicline-Adjunctive-Treatment-in-Schizophrenia.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline: Varenicline Treatment Group
- Placebo: Placebo Control Group
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 35 | 34
Week 2 | 32 | 33
Week 8 | 32 | 27
Completed | 32 | 27
Not Completed | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Continuous [Mean (Standard Deviation); unit: years]
  Smoker | 43.0 (2.5) | 41.5 (2.5) | 42.2 (2.5)
  Non-Smoker | 45.7 (2.6) | 42.1 (3.2) | 43.9 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline data were available for participants who completed 2 weeks in the study
  Participants
    Female | 12 | 10 | 22
    Male | 23 | 24 | 47
Region of Enrollment [Number; unit: participants]
  United States | 35 | 34 | 69
BPRS Total [Mean (Standard Deviation); unit: units on a scale] — BRIEF PSYCHIATRIC RATING SCALE has 20 items:
  1 = not present, 2 = very mild, 3 = mild, 4 = moderate, 5 = moderately severe, 6 = severe, 7 = extremely severe. Score range from 20 to 140.
  units on a scale
    Smoker | 36.2 (1.9) | 35.0 (2.0) | 35.6 (1.9)
    Non-Smoker | 31.2 (2.0) | 34.0 (2.5) | 32.6 (2.2)
Ham-D Total Score [Mean (Standard Deviation); unit: units on a scale] — HAMILTON DEPRESSION RATING SCALE In general, the higher the total score the more severe the depression. One can use the following to classify severity: 0 - 13 mild; 14-17 mild to moderate; >17 moderate to severe. However, in this trial, these categorical classifications of severity were not used. Only the raw score was used to compare between the treatment arm and the placebo arm.
  units on a scale
    Smoker | 5.0 (0.9) | 5.76 (1.15) | 5.38 (1.0)
    Nonsmoker | 5.2 (0.7) | 6.6 (1.0) | 5.8 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (Ham-D)
Description: Ham-D Total Score (range 0 to 54, higher score is worse). Definition is fully described in a peer-review journal reported at Arch Gen Psychiatry 2011 Dec;68(12):1195-206.
Time Frame: Week 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 32 | 27
units on a scale
  Smoker | 22.9 (3.2) | 20.6 (3.4)
  Nonsmoker | 19.4 (3.2) | 18.6 (2.2)

2. Primary Outcome: Memory Saccadic Positional Error, Degrees
Description: A saccade is a quick eye movement. Spatial working memory was assessed by memory saccade. Participants were asked to focus on a target while a peripheral cue was flashed. Participants were signaled to look in the direction of the peripheral cue when the central target was removed, and the positional error was calculated as the distance between the saccadic and peripheral target positions. Definition is fully described in a peer-review journal reported at Arch Gen Psychiatry 2011 Dec;68(12):1195-206.
Time Frame: Week 8
Measure: Mean (Standard Error); unit: degrees
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 32 | 27
degrees
  Smoker | 1.6 (0.2) | 1.7 (0.2)
  Nonsmoker | 1.7 (0.1) | 1.8 (0.2)

3. Primary Outcome: Predictive Pursuit Gain
Description: Pursuit gain is the averaged artifact-free eye velocity divided by target velocity. Participants are asked to track a target with their eyes. Participants may use a predictive mechanism to perform the tracking. The pursuit gain using the predictive mechanism is calculated. Further definition is fully described in a peer-review journal reported at Arch Gen Psychiatry 2011 Dec;68(12):1195-206.
Time Frame: Week 8
Measure: Mean (Standard Error); unit: velocity ratio
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 32 | 27
velocity ratio
  Smoker | 0.31 (0.03) | 0.34 (0.04)
  Nonsmoker | 0.24 (0.04) | 0.31 (0.04)

4. Primary Outcome: Maintenance Pursuit Gain
Description: Pursuit gain is the averaged artifact-free eye velocity divided by target velocity. Eye velocity during the regular eye-tracking period (without foveal stabilization) divided by target velocity was used to calculate the maintenance pursuit gain. Further definition is fully described in a peer-review journal reported at Arch Gen Psychiatry 2011 Dec;68(12):1195-206.
Time Frame: Week 8
Measure: Mean (Standard Error); unit: velocity ratio
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 32 | 27
velocity ratio
  Smoker | 0.8 (0.1) | 0.8 (0.04)
  Nonsmoker | 0.8 (0.1) | 0.8 (0.1)

5. Primary Outcome: Digit Symbol Test
Description: Digit symbol test score (0 to no definite upper range, higher score is better). Definition is fully described in a peer-review journal reported at Arch Gen Psychiatry 2011 Dec;68(12):1195-206.
Time Frame: Week 0, Week 2 and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Varenicline: Varenicline
  Varenicline: Varenicline 0.5mg po qd x 7 days then titrated to Varenicline 0.5mg po bid x 7 weeks
- Placebo: Placebo
  Placebo: Placebo 0.5mg po qd x 7 days then titrated to Placebo 0.5mg po bid x 7 weeks
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 28 | 28
units on a scale
  Week 0 | 53.9 (19.3) | 53.2 (19.1)
  Week 2 | 55.9 (19.0) | 53.8 (20.6)
  Week 8 | 54.2 (20.3) | 54.3 (21.7)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Mixed model ANCOVA in which baseline served as the covariate and Smoking status and measurement occasions were between and within-groups factors, respectively; Test type: Superiority or Other; p < 0.05, ANCOVA

6. Primary Outcome: Conner's Continuous Performance Test (CPT) Detectability Score
Description: Conner's CPT Detectability Score (no set normal range, higher is generally better). Definition is fully described in a peer-review journal reported at Arch Gen Psychiatry 2011 Dec;68(12):1195-206.
Time Frame: Week 0, Week 2 and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Varenicline: Varenicline
- Placebo: Placebo
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 30 | 26
units on a scale
  Week 0 | 0.87 (0.38) | 0.87 (0.50)
  Week 2 | 0.89 (0.42) | 0.97 (0.54)
  Week 8 | 0.95 (0.48) | 0.97 (0.53)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Mixed model ANCOVA in which baseline CPT Detectability served as the covariate and Smoking status and measurement occasions were between and within-groups factors, respectively; Test type: Superiority or Other; p > 0.05, ANCOVA — All treatment main and interaction effect p-values were > 0.05

7. Primary Outcome: Antisaccade Error Rates
Description: In antisaccade, participants were asked to focus on a central target. When a peripheral cue was presented, participants were asked to look in an equidistant and opposite direction of the peripheral cue. The error rate is calculated as the number of trials in which the participant looked toward the cue, rather than in the opposite direction, divided by the total number of trials. Further definition is fully described in a peer-review journal reported at Arch Gen Psychiatry 2011 Dec;68(12):1195-206.
Time Frame: Week 0, Week 2 and Week 8
Measure: Mean (Standard Deviation); unit: percentage errors
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 31 | 27
percentage errors
  Week 0 | 0.61 (0.27) | 0.54 (0.27)
  Week 2 | 0.49 (0.27) | 0.54 (0.26)
  Week 8 | 0.45 (0.26) | 0.53 (0.28)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Mixed model ANCOVA in which baseline Antisaccade Errors served as the covariate and Smoking status and measurement occasions were between and within-groups factors, respectively; Test type: Superiority or Other; p < 0.05, ANCOVA

8. Primary Outcome: P50
Description: P50 response is a measure of the amplitude of the brain wave in response to a sound, where the positive going amplitude of the brain wave occurring at about 50 milliseconds after the sound. Further definition is fully described in a peer-review journal reported at Arch Gen Psychiatry 2011 Dec;68(12):1195-206.
Time Frame: Week 0, Week 2 and Week 8
Measure: Mean (Standard Error); unit: microvolts
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 31 | 32
microvolts
  Week 0 | 3.2 (0.73) | 3.1 (.71)
  Week 2 | 3.2 (0.75) | 3.0 (.72)
  Week 8 | 3.2 (0.6) | 2.5 (.77)

ADVERSE EVENTS:
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 0/35 | 0/34

LIMITATIONS AND CAVEATS:
The small number of nonsmokers in the placebo arm could have led to reduced power and false negatives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes